CLINICAL TRIAL: NCT04156776
Title: Comparison Of Muscle Energy Technique And Active Isolated Stretching On Erector Spinae Muscle In The Management Of Mechanical Low Back Pain
Brief Title: Comparison of MET and AIS on Erector Spinae Muscle in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Hanan Zafar-REC/00387
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Mechanical Low Back Pain
Keywords: Active Isolated Stretching; Muscle Energy Technique; Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Group A (MET) and Group B (AIS)
Who Masked: Participant
Masking Description: Patients were not aware about the groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (MET) (Experimental): Muscle Energy Technique Conventional Treatment
  Interventions: Other: Muscle Energy Technique; Other: Conventional Treatment
- Group B (AIS) (Experimental): Active Isolated Stretching Conventional Treatment
  Interventions: Other: Active Isolated Stretching; Other: Conventional Treatment

INTERVENTIONS:
Other: Muscle Energy Technique — Muscle energy technique was repeated 4 times per session every day for 3 days a week for 4 weeks after the application of moist heating pad for 30 minutes before each session.
  Arms: Group A (MET)
Other: Active Isolated Stretching — The patient was asked to sit in an upright seated position and flex his/her knees 12 to 18 inches. Patient was asked to tuck the chin, exhale, and firmly contract the abdominal muscles as he/she curls their body forward. He/she was also guided not to bounce or make rapid movements at the end range of the active motion. Then, he was asked to move back to the starting position and repeat the same procedure for 8 to 10 times. Stretch on the end range was not more than 2 seconds.
  This technique was repeated 10 times per session every day for 3 days a week for 4 weeks after the application of moist heating pad for 30 minutes before each session.
  Arms: Group B (AIS)
Other: Conventional Treatment — Conventional physical therapy treatment includes the application of moist heating pad for 30 minutes on lower back/ lumbar region prior to the intervention to both groups.

SUMMARY:
The main objective of the study was to compare the effectiveness of Muscle Energy Technique and Active Isolated Stretching on Erector Spinae Muscle in the management of Mechanical Low back Pain (LBP) and to find out that which technique is better for the treatment of mechanical LBP

DETAILED DESCRIPTION:
Lumbar spine "mobilization and manipulation" relieves the hypomobility in the intervertebral joints which results in pain reduction and significant improvement in lumbar spine ROMs. In dry needling, trigger point is palpated and tiny needle is inserted in hyperirritable point. Local twitch response is noted. Referred pain pattern may appear followed by pain relief and trigger point release. In this technique, pain is relieved by spontaneous positioning and maintains a non-painful tension in hypertonic muscle. When subject is placed in a non-tension position pain is decreased up to 70%. In Instrument assisted soft tissue mobilization: Various instruments like beveled edges,tools are used for soft tissue mobilization and decreasing pain threshold.

MUSCLE ENERGY TECHNIQUE (MET) is actually a sort of "myofascial release soft-tissue method" in which the patient is given a command to use the muscles actively in a direction opposite to the force applied by the therapist which results in the enhancement of joint ROM and flexibility. In MET, "sub-maximal active resisted isometric contraction of muscle" is performed for couple of times after that the muscle is stretched passively which results in the increment in ROM, desired muscular length and flexibility.

The concept which is used in MET is the reciprocal inhibition in which "the muscle which is faulty placed in mid range and the practitioner resists the greatest power either isotonically or isometrically". The patient is instructed to breathe in with the application of force and breathe out as the muscle is being lengthened For convenience, therapeutic exercises and specialized manual therapy treatment protocols can be divided into two main levels although the treatment of LBP depends on the condition of patient, intensity of pain, diagnosis and signs and symptoms. First level includes therapeutic exercises like "Range of Motion (ROM) exercises, stretching exercises, strengthening exercises and aerobic exercises" whereas second level includes advances manual therapy treatment protocols which includes specialised techniques like dry needling, strain counter strain, , lumbar stabilization exercises, MET, AIS etc When patient performs the exercises actively, nutritional supply gets enhanced to the soft tissues in lower back which keeps the vertebras, muscles, joints and ligaments sound. Lower back exercises keep the patient's spine healthy by maintaining its flexibility and strength and additionally, they decrease the chances of re-occurrence of LBP.

Most commonly advised back exercises by physical therapists in the management of low back pain are "aerobic conditioning, stretching exercises, and strengthening exercises, McKenzie Exercises and lumbar stabilization exercises Lower back stretching exercises increase ROM and improves flexibility. Literature also recommends to stretch "hamstrings, piriformis and gluteal muscles" once or twice a day. Stretching exercises includes hamstring stretch or straight leg raising (SLR), knee to chest stretch, piriformis muscle stretch, etc Lower back stretching exercises increase ROM and improves flexibility. Literature also recommends to stretch "hamstrings, piriformis and gluteal muscles" once or twice a day. Stretching exercises includes hamstring stretch or SLR, knee to chest stretch, piriformis muscle stretch, etc On alternate days, doing aerobic exercises for 30 to 40 minutes a day for three times in a week, helps in the long-term reduction of LBP because by these exercises, nutrition supply can be enhanced to the soft tissues which promotes healing. Such type of exercises includes "walking, jogging, bicycling, swimming, etc Mobilization of lumbar spine, electrotherapy treatment, Stretching and strengthening exercises, postural correction of the individuals which are suffering from LBP are routine treatment protocols. Conventional physical therapy treatment is effective as it decreases the pain and improves the patient's functional outcome for patients of chronic LBP, but erector spinae muscle length remains compromised. Muscle energy technique and Active isolated stretching technique are advanced treatment protocols for getting improvement in muscle length by which patients get better in few sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients having acute mechanical LBP.
* Patients having restricted ROM.

Exclusion Criteria:

* Patients with ankylosing spondylitis.
* Patient undergone any spinal surgery.
* Patient having scoliosis.
* Patient with tumor.
* Patient with Rheumatoid Arthritis and other systemic diseases.
* Immobile/ Bed ridden patients.
* Patients with cognitive Problems. 8. Patients having vertebral compression fracture. 9. Patients with slump test positive.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Erector Spinae Muscle Length through Measuring Tape | 4th week
  The length of the erector spinae can be evaluated in seated position with the legs fully flexed off the end of the table. The therapist stands behind the patient and palpates the anterior superior iliac spine (ASIS) bilaterally. The patient was taught and instructed to perform a posterior pelvic tilt, thus flattening the lumbar lordosis by creating lumbar flexion. Then, the patient was instructed to flex forward, attempting to bring the forehead to the knees. The practitioner feels for when the ASIS of the patient begins to move, which would indicate the end of thoracolumbar flexion and would indicate the initiation of an anterior pelvic tilt.
  Patient's forehead should come within 10 inches of the knees. The therapist had to note that no knee flexion occurred and the movement is coming from the thoracolumbar spine only.
  In the current study, erector spinae muscle length was measured prior starting the treatment as well as after completing the last treatment session.
Oswestry Disability Index (ODI) | 4th week
  ODI is the tool to measure the level of disability in essential conditions. This scale totally focuses on the evaluation of disability and impairment caused due to LBP. It contains 10 questions which are easily understandable. The very first question in the questionnaire is about the intensity of pain while next questions are about the level of disability and impairment caused on activity of daily living (ADLs) which includes "sleep, lifting, walking, sex life, sitting and so forth." Score for each question is from zero, which indicates no intensity, to five which indicates greatest inability due to LBP. Total obtained score of ten questions was calculated which was divided by the total possible score (i.e., 50) and then it was multiplied by hundred. The answer was in percentage. Let's assume, the total score of the patient was 20 and total possible score is 50 then 20/50 x 100 = 40 %.
Numeric Pain Rating Scale (NPRS) | 4th week
  NPRS is a tool to measure the pain intensity. Frequently, pain is the main concern of the patient which compelled him/ her to pursue treatment and NPRS is essential tool to gauge pain intensity in routine practice although psychological aspects of pain can also be considered. NPRS contains eleven levels from zero, which presents "no pain", till ten which presents the "worst pain" one can feel, as shown in figure 11. NPRS is an exceptionally easy to quantify pain, can be used by the patient him self and even it can likewise be utilized in people with low proficiency. It is utilized routinely in numerous nations and languages.

SECONDARY OUTCOMES:
Lumbar Spine ROM through Inclinometer | 4th week
  Lumbar spine range of motion was performed in standing position with help of "inclinometer". The "American Medical Association" issued the guidelines in which the use of inclinometers has been declared as "a feasible and potentially accurate method of measuring spine mobility." In current study, dual- inclinometer method was used to measure the lumbar spine ROM of "flexion, extension, right and left side bending" prior starting the treatment as well as after completing the last treatment session. Diseases of lumbar spine, spinal muscular issues reduce the lumbar spine ROM. ROM values for normal lumbar spine.
  Patient was in standing position. Baseline inclinometer was placed on the "midline of spine in line with Posterior superior iliac spine (PSIS)" and superior inclinometer was placed "15 cm above baseline landmark". Patient was asked to flex the spine as much as he/she can. Inclinometers was placed in above mentioned points by the therapist till the end of possible ROM.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali, S., et al., CHRONIC LOW BACK PAIN; EFFECTS OF THE LUMBAR STABILIZATION EXERCISES ON PAIN, RANGE OF MOTION AND FUNCTIONAL DISABILITY IN THE MANAGEMENT. Professional Medical Journal, 2017. 24(4).
- [Background] Lawrence RC, Helmick CG, Arnett FC, Deyo RA, Felson DT, Giannini EH, Heyse SP, Hirsch R, Hochberg MC, Hunder GG, Liang MH, Pillemer SR, Steen VD, Wolfe F. Estimates of the prevalence of arthritis and selected musculoskeletal disorders in the United States. Arthritis Rheum. 1998 May;41(5):778-99. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-V. PMID 9588729
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Hoy D, March L, Brooks P, Woolf A, Blyth F, Vos T, Buchbinder R. Measuring the global burden of low back pain. Best Pract Res Clin Rheumatol. 2010 Apr;24(2):155-65. doi: 10.1016/j.berh.2009.11.002. PMID 20227638
- [Background] Chien JJ, Bajwa ZH. What is mechanical back pain and how best to treat it? Curr Pain Headache Rep. 2008 Dec;12(6):406-11. doi: 10.1007/s11916-008-0069-3. PMID 18973732
- [Background] Endean A, Palmer KT, Coggon D. Potential of magnetic resonance imaging findings to refine case definition for mechanical low back pain in epidemiological studies: a systematic review. Spine (Phila Pa 1976). 2011 Jan 15;36(2):160-9. doi: 10.1097/BRS.0b013e3181cd9adb. PMID 20739918
- [Background] Linton SJ. The relationship between activity and chronic back pain. Pain. 1985 Mar;21(3):289-294. doi: 10.1016/0304-3959(85)90092-2. PMID 3157914
- [Background] Okunribido OO, Magnusson M, Pope MH. The role of whole body vibration, posture and manual materials handling as risk factors for low back pain in occupational drivers. Ergonomics. 2008 Mar;51(3):308-29. doi: 10.1080/00140130701637262. PMID 18311609
- [Background] Drake, R., A.W. Vogl, and A.W. Mitchell, Gray's Anatomy for Students E-Book. 2009: Elsevier Health Sciences
- [Background] Galbusera, F. and H.-J. Wilke, Biomechanics of the Spine: Basic Concepts, Spinal Disorders and Treatments. 2018: Academic Press
- [Background] Frankel VH. Biomechanics of the musculoskeletal system. Introduction. Arch Surg. 1973 Sep;107(3):405. doi: 10.1001/archsurg.1973.01350210041013. No abstract available. PMID 4783034
- [Background] Adrian, M. and J.M. Cooper, Biomechanics of human movement. 1995: Brown & Benchmark
- [Background] Kaltenborn, F.M., et al., Manual Mobilization of the Joints: The Spine. 2009: Orthopedic Physical Therapy
- [Background] Cramer, G.D. and S.A. Darby, Clinical Anatomy of the Spine, Spinal Cord, and ANS. 2017: Elsevier Health Sciences
- [Background] Hans, J., D. Kachlík, and R.S. Tubbs, An Illustrated Terminologia Neuroanatomica: A Concise Encyclopedia of Human Neuroanatomy. 2018: Springer
- [Background] Roth R, Donath L, Kurz E, Zahner L, Faude O. Absolute and relative reliability of isokinetic and isometric trunk strength testing using the IsoMed-2000 dynamometer. Phys Ther Sport. 2017 Mar;24:26-31. doi: 10.1016/j.ptsp.2016.11.005. Epub 2016 Nov 30. PMID 27964928
- [Background] Gill C, Sanford J, Binkley J, Stratford P, Finch E. Low back pain: program description and outcome in a case series. J Orthop Sports Phys Ther. 1994 Jul;20(1):11-6. doi: 10.2519/jospt.1994.20.1.11. PMID 8081403
- [Background] Gupta, B., Spondylosis: A Scientometric Assessment of Global Publications Output during 2008-17. EC Orthopaedics, 2018. 9: p. 331-339
- [Background] Weinstein, P.R., G. Ehni, and C.B. Wilson, Lumbar Spondylosis: Diagnosis, Management, and Surgical Treatment. 1977: Year Book Medical Publishers
- [Background] Weisman, M.H., J.D. Reveille, and D. van der Heijde, Ankylosing Spondylitis and the Spondyloarthropathies. 2006: Mosby/Elsevier
- [Background] Gunzburg, R. and M. Szpalski, Lumbar Spinal Stenosis. 2000: Lippincott Williams & Wilkins
- [Background] Gunzburg, R. and M. Szpalski, Lumbar Disk Herniation. 2002: Lippincott Williams & Wilkins
- [Background] Anderson, G., The epidemiology of spinal disorders. The adult spine: principles and practice, 1997
- [Background] Krause N, Ragland DR. Occupational disability due to low back pain: a new interdisciplinary classification based on a phase model of disability. Spine (Phila Pa 1976). 1994 May 1;19(9):1011-20. doi: 10.1097/00007632-199405000-00002. PMID 8029734
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Manusov EG. Evaluation and diagnosis of low back pain. Prim Care. 2012 Sep;39(3):471-9. doi: 10.1016/j.pop.2012.06.003. PMID 22958556
- [Background] Deyo RA, Diehl AK, Rosenthal M. How many days of bed rest for acute low back pain? A randomized clinical trial. N Engl J Med. 1986 Oct 23;315(17):1064-70. doi: 10.1056/NEJM198610233151705. PMID 2945109
- [Background] van Tulder M, Becker A, Bekkering T, Breen A, del Real MT, Hutchinson A, Koes B, Laerum E, Malmivaara A; COST B13 Working Group on Guidelines for the Management of Acute Low Back Pain in Primary Care. Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S169-91. doi: 10.1007/s00586-006-1071-2. No abstract available. PMID 16550447
- [Background] Burnett MG, Stein SC, Bartels RH. Cost-effectiveness of current treatment strategies for lumbar spinal stenosis: nonsurgical care, laminectomy, and X-STOP. J Neurosurg Spine. 2010 Jul;13(1):39-46. doi: 10.3171/2010.3.SPINE09552. PMID 20594016
- [Background] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Background] Hansen FR, Bendix T, Skov P, Jensen CV, Kristensen JH, Krohn L, Schioeler H. Intensive, dynamic back-muscle exercises, conventional physiotherapy, or placebo-control treatment of low-back pain. A randomized, observer-blind trial. Spine (Phila Pa 1976). 1993 Jan;18(1):98-108. doi: 10.1097/00007632-199301000-00015. PMID 8434332
- [Background] French SD, Cameron M, Walker BF, Reggars JW, Esterman AJ. A Cochrane review of superficial heat or cold for low back pain. Spine (Phila Pa 1976). 2006 Apr 20;31(9):998-1006. doi: 10.1097/01.brs.0000214881.10814.64. PMID 16641776
- [Background] Marchand S, Charest J, Li J, Chenard JR, Lavignolle B, Laurencelle L. Is TENS purely a placebo effect? A controlled study on chronic low back pain. Pain. 1993 Jul;54(1):99-106. doi: 10.1016/0304-3959(93)90104-W. PMID 8378107
- [Background] van der Windt DAWM, van der Heijden GJMG, van den Berg SGM, Ter Riet G, de Winter AF, Bouter LM. Ultrasound therapy for musculoskeletal disorders: a systematic review. Pain. 1999 Jun;81(3):257-271. doi: 10.1016/S0304-3959(99)00016-0. PMID 10431713
- [Background] Franca FR, Burke TN, Hanada ES, Marques AP. Segmental stabilization and muscular strengthening in chronic low back pain: a comparative study. Clinics (Sao Paulo). 2010;65(10):1013-7. doi: 10.1590/s1807-59322010001000015. PMID 21120303
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Lewis, C. and T.W. Flynn, The use of strain-counterstrain in the treatment of patients with low back pain. Journal of Manual & Manipulative Therapy, 2001. 9(2): p. 92-98.
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Sherman KJ, Cherkin DC, Wellman RD, Cook AJ, Hawkes RJ, Delaney K, Deyo RA. A randomized trial comparing yoga, stretching, and a self-care book for chronic low back pain. Arch Intern Med. 2011 Dec 12;171(22):2019-26. doi: 10.1001/archinternmed.2011.524. Epub 2011 Oct 24. PMID 22025101
- [Background] Risch SV, Norvell NK, Pollock ML, Risch ED, Langer H, Fulton M, Graves JE, Leggett SH. Lumbar strengthening in chronic low back pain patients. Physiologic and psychological benefits. Spine (Phila Pa 1976). 1993 Feb;18(2):232-8. PMID 8185727
- [Background] Sculco AD, Paup DC, Fernhall B, Sculco MJ. Effects of aerobic exercise on low back pain patients in treatment. Spine J. 2001 Mar-Apr;1(2):95-101. doi: 10.1016/s1529-9430(01)00026-2. PMID 14588388
- [Background] Koes BW, Assendelft WJ, van der Heijden GJ, Bouter LM. Spinal manipulation for low back pain. An updated systematic review of randomized clinical trials. Spine (Phila Pa 1976). 1996 Dec 15;21(24):2860-71; discussion 2872-3. doi: 10.1097/00007632-199612150-00013. PMID 9112710
- [Background] Bronfort G, Haas M, Evans RL, Bouter LM. Efficacy of spinal manipulation and mobilization for low back pain and neck pain: a systematic review and best evidence synthesis. Spine J. 2004 May-Jun;4(3):335-56. doi: 10.1016/j.spinee.2003.06.002. PMID 15125860
- [Background] Simons DG, Travell JG. Myofascial origins of low back pain. 1. Principles of diagnosis and treatment. Postgrad Med. 1983 Feb;73(2):66, 68-70, 73 passim. doi: 10.1080/00325481.1983.11697756. PMID 6218489
- [Background] Yuan QL, Guo TM, Liu L, Sun F, Zhang YG. Traditional Chinese medicine for neck pain and low back pain: a systematic review and meta-analysis. PLoS One. 2015 Feb 24;10(2):e0117146. doi: 10.1371/journal.pone.0117146. eCollection 2015. PMID 25710765
- [Background] Hammer, W.I., Functional soft-tissue examination and treatment by manual methods. 2007: Jones & Bartlett Learning.
- [Background] Frank, C., P. Page, and R. Lardner, Assessment and treatment of muscle imbalance: the Janda approach. 2009: Human kinetics.
- [Background] Chaitow, L. and K. Crenshaw, Muscle energy techniques. 2006: Elsevier Health Sciences.
- [Background] Page P. Current concepts in muscle stretching for exercise and rehabilitation. Int J Sports Phys Ther. 2012 Feb;7(1):109-19. PMID 22319684
- [Background] Lenehan, K.L., G. Fryer, and P. McLaughlin, The effect of muscle energy technique on gross trunk range of motion. Journal of osteopathic medicine, 2003. 6(1): p. 13-18.
- [Background] Wilson E, Payton O, Donegan-Shoaf L, Dec K. Muscle energy technique in patients with acute low back pain: a pilot clinical trial. J Orthop Sports Phys Ther. 2003 Sep;33(9):502-12. doi: 10.2519/jospt.2003.33.9.502. PMID 14524509
- [Background] Selkow NM, Grindstaff TL, Cross KM, Pugh K, Hertel J, Saliba S. Short-term effect of muscle energy technique on pain in individuals with non-specific lumbopelvic pain: a pilot study. J Man Manip Ther. 2009;17(1):E14-8. doi: 10.1179/jmt.2009.17.1.14E. PMID 20046557
- [Background] Mattes, A.L., Active isolated stretching. Journal of Bodywork and Movement Therapies, 1996. 1(1): p. 28-33.
- [Background] Mattes, A.L., Active isolated stretching: the Mattes method. 2000: AL Mattes
- [Background] Bernhart, C.M., A review of stretching techniques and their effects on exercise. 2013.
- [Background] Liemohn, W., N. Mazis, and S. Zhang, Effect Of Active Isolated And Static Stretch Training On Active Straight Leg Raise Performance. Medicine & Science in Sports & Exercise, 1999. 31(5): p. S116.
- [Background] Thakur, A., Running economy: Acute effect of active isolated stretching. 2009: Lamar University-Beaumont.
- [Background] Ellythy, M.A., Efficacy of Muscle Energy Technique Versus Strain Counter Strain on Low Back Dysfunction. Bulletin of Faculty of Physical Therapy, 2012. 17(2).
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Berryman, R.N. and W.D. Bandy, Joint range of motion and muscle length testing. Missouri: Elsevier, 2010.
- [Background] Funk D, Swank AM, Adams KJ, Treolo D. Efficacy of moist heat pack application over static stretching on hamstring flexibility. J Strength Cond Res. 2001 Feb;15(1):123-6. PMID 11708695
- [Background] Joshi, R., et al., Effect of Muscle Energy Technique on Pain And Function in Patients With Sacroiliac Dysfunction-Experimental Study. International Journal Of Scientific Research And Education, 2017. 5(06).
- [Background] Balani, S. and C. Kataria, Comparing Effectiveness of Suboccipital Muscle Energy Technique Alone, Passive Hamstring Stretching Technique Alone and Combination of both for Improving Hamstring Muscle Flexibility in Healthy Collegiate Subjects. Int J Heal Sci Res, 2015. 5(8): p. 329-336.
- [Background] El-Bandrawy, A.M., M.A. Mohamed, and A.M. Mamdouh, Effect of Muscle Energy Technique on Pain Perception and Functional Disability of Women with Postnatal Low Back Pain. British Journal of Medicine and Medical Research, 2014. 4(33): p. 5253.
- [Background] Abutaleb, E.E., M.T. Eldesoky, and S.A. El Rasol, Effect of Muscle Energy Technique on Anterior Pelvic Tilt in Lumbar Spondylosis Patients. World Academy of Science, Engineering and Technology, International Journal of Medical, Health, Biomedical, Bioengineering and Pharmaceutical Engineering, 2015. 9(8): p. 651-655.
- [Background] Middag, T.R. and P. Harmer, Active-isolated stretching is not more effective than static stretching for increasing hamstring ROM. Medicine & Science in Sports & Exercise, 2002. 34(5): p. S151.